CLINICAL TRIAL: NCT07176468
Title: Efficacy of Personalized iTBS in Real-World Clinical Settings for Alleviating Schizophrenia Symptoms : A Randomized Single-Blind Trial
Brief Title: Personalized iTBS in Real-World Clinical Settings for Schizophrenia
Acronym: EPSREAL-SC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head of the Department, Department of Neurology, The First Affiliated Hospital of Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHMU-SCZ-RWTBS
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Transcranial Magnetic Stimulation
Keywords: schizophrenia; transcranial magnetic stimulation; Functional Magnetic Resonance Imaging (fMRI)
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:Neuronavigation-guided individualized intermittent theta burst stimulation (iTBS) (Experimental): Participants will receive iTBS daily for 2 week within real-world treatment settings
  Interventions: Other: Neuronavigation-guided individualized iTBS
- Control group: ordinary drug treatment (No Intervention): The participants will receive regular medication treatment every day for 2 week.

INTERVENTIONS:
Other: Neuronavigation-guided individualized iTBS — Participants will receive individualized iTBS for 14 consecutive days in addition to their usual medication regimen.
  iTBS parameters: 50 Hz bursts every 200 ms (5 Hz), 2s on/8s off, total 600 pulses per session;6 sessions/day (3 in morning, 3 in afternoon, 3600 pulses/day); 100% RMT intensity; Neuronavigation: Brainsight system (Rogue Research, Canada)
  Other Names: iTBS
  Arms: Experimental:Neuronavigation-guided individualized intermittent theta burst stimulation (iTBS)

SUMMARY:
This study is designed to determine whether neuronavigation-guided, personalized Intermittent Theta-Burst Stimulation (iTBS) can produce clinically benefits for patients with schizophrenia when delivered in real-world treatment settings. By situating the intervention within real-world treatment settings-without imposing restrictions on concurrent pharmacotherapy-this trial seeks to generate evidence that is both scientifically rigorous and clinically relevant.

The main questions it seeks to address are:

Does the personalized iTBS target TMS protocol improve clinical symptoms in patients with schizophrenia within real-world treatment settings? What neural circuit changes, as assessed by functional MRI, occur following TMS treatment?

Participants will:

Undergo personalized,personalized iTBS target treatment daily for 2 weeks. Complete baseline and post-treatment assessments, including clinical symptom scales (PANSS, HAMA, HAMD) and neuropsychological tests (MoCA, DST, VFT, Stroop Test, and AVLT).

Have structural and resting-state functional MRI scans before and after treatment.

Be monitored for any treatment-related adverse events.

DETAILED DESCRIPTION:
Effective intervention is critical for reducing relapse risk, improving long-term prognosis, and lowering healthcare costs for schizophrenia.The present study therefore aims to assess whether neuronavigation-guided, individualized Intermittent Theta-Burst Stimulation (iTBS) can accelerate symptom improvement in schizophrenia when delivered in real-world clinical settings. By situating the intervention within real-world treatment settings-without imposing restrictions on concurrent pharmacotherapy-this trial seeks to generate evidence that is both scientifically rigorous and clinically relevant. Patients with schizophrenia will be prospectively recruited and received 2 weeks of iTBS treatment.

Before treatment, structural and resting-state functional MRI data wil be collected from each patient. Clinical symptom severity will be assessed using the Positive and Negative Syndrome Scale (PANSS), Hamilton Anxiety Rating Scale (HAMA), and Hamilton Depression Rating Scale (HAMD). For patients experiencing auditory verbal hallucinations, the Auditory Hallucination Rating Scale (AHRS) will be also administered. Additionally, a battery of neuropsychological tests will be conducted, including the Montreal Cognitive Assessment (MoCA), Digit Span Test (DST), Verbal Fluency Test (VFT), Stroop Test, and Chinese Auditory Verbal Learning Test (AVLT).

After completing the 2-week iTBS treatment, clinical symptom severity, treatment-related adverse events wil be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years, any gender
* Meets DSM-5 criteria for schizophrenia
* Antipsychotic medication change (initiation, dose adjustment, or switch) occurred within the past 3 days
* Capable of understanding the study and providing written informed consent Able to comply with study procedures and complete assessments

Exclusion Criteria:

* Active suicidal ideation or behavior
* Major neurological disorders (e.g., epilepsy, organic brain lesions, severe head trauma)
* Contraindications to MRI or TMS (e.g., metal implants, pacemakers)
* Pregnancy or lactation
* Receipt of TMS or ECT within the past 6 months
* Judged by investigators to be unsuitable for participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
The Positive and Negative Syndrome Scale (PANSS) | baseline and week 2 (post-treatment)
  The primary outcome was the changes in the Positive and Negative Syndrome Scale (PANSS) total scores from baseline to week 2. PANSS total score range 30 to 210, the higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) subscales | baseline and week 2 (post-treatment)
  Secondary outcomes included changes in the PANSS subscales score. PANSS positive score and negative score range 7 to 49, the higher scores indicate more severe symptoms. PANSS general score range 16 to 112, the higher scores indicate more severe symptoms.
Hamilton Anxiety Rating Scale (HAMA) | baseline and week 2 (post-treatment)
  Secondary outcomes included changes in the HAMA score. HAMA scale scores range from 0 to 56 points, the higher the score indicates the more serious anxiety
Hamilton Depression Rating Scale (HAMD) | baseline and week 2 (post-treatment)
  Secondary outcomes included changes in the HAMD score. HAMA scale scores range from 0 to 50 points, the higher the score indicates the more serious depression.
Auditory Hallucination Rating Scale (AHRS) | baseline and week 2 (post-treatment)
  The changes in the Auditory Hallucination Rating Scale (AHRS) score were also included as a secondary outcome. AHRS range 0 to 41, the higher scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No